CLINICAL TRIAL: NCT02651584
Title: A Phase III, Randomized, Double-Blind, Active-Controlled, Parallel Group, Multi-center Trial Assessing the Efficacy and Safety of a Once-Weekly and Once-Monthly, Long-Acting Subcutaneous Injectable Depot of Buprenorphine (CAM2038) in Treatment of Adult Outpatients With Opioid Use Disorder
Brief Title: Clinical Trial of CAM2038, Long-acting Subcutaneous Buprenorphine Injections for Treatment of Patients With Opioid Dependence
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Braeburn Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HS-11-421
Record Dates: First submitted 2015-12-30; First posted 2016-01-11 (Estimated); Results first posted 2019-08-22 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2018-08

CONDITIONS: Opioid Use Disorders
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine; Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SL BPN/NX tabs + placebo SC injections (Experimental): SL BPN/NX: 2 mg/0.5 mg or 8 mg/2 mg BPN/naloxone tablets administered daily, at doses of 8 mg/2 mg to 32 mg/8 mg per day.
  CAM2038 placebo: 0.16, 0.32, 0.48 and 0.64 mL SC injection administered once weekly or once monthly (matching volumes for CAM2038 q1w and near-matching volumes for CAM2038 q4w).
  Interventions: Drug: SL BPN/NX tabs; Drug: placebo SC injections
- CAM2038 SC injections + SL placebo tabs (Experimental): CAM2038 q1w: BPN FluidCrystal® SC injection depot for once weekly administration (50 mg/mL) at doses of 8, 16, 24 or 32 mg (BPN base) (0.16, 0.32, 0.48 or 0.64 mL SC injection).
  CAM2038 q4w: BPN FluidCrystal® SC injection depot for once monthly administration (356 mg/mL) at doses of 64, 96, 128 or 160 mg (BPN base) (0.18, 0.27, 0.36 or 0.45 mL SC injection).
  SL placebo: tablets matching 2 mg/0.5 mg and 8 mg/2 mg SL BPN doses, administered daily
  Interventions: Drug: CAM2038 SC injection; Drug: SL placebo tablets

INTERVENTIONS:
Drug: CAM2038 SC injection
  Other Names: Buprenorphine injection
  Arms: CAM2038 SC injections + SL placebo tabs
Drug: SL BPN/NX tabs
  Other Names: Suboxone
  Arms: SL BPN/NX tabs + placebo SC injections
Drug: placebo SC injections
  Other Names: placebo
  Arms: SL BPN/NX tabs + placebo SC injections
Drug: SL placebo tablets
  Other Names: placebo
  Arms: CAM2038 SC injections + SL placebo tabs

SUMMARY:
Phase III, randomized, double-blind, double-dummy, active-controlled, parallel group multi-center trial, designed to evaluate the non-inferiority of CAM2038 compared to an existing standard of care (SL BPN/NX) in initiation and maintenance treatment with BPN.

DETAILED DESCRIPTION:
This is a Phase III, randomized, double-blind, double-dummy, active-controlled, parallel group multi-center trial, designed to evaluate the non-inferiority of CAM2038 compared to an existing standard of care (SL BPN/NX) in initiation and maintenance treatment with BPN. The trial will involve 4 phases: Screening, Phase 1 (weekly visits), Phase 2 (monthly visits), and Follow-up.

Approximately 380 subjects (190 subjects per arm) will be randomized.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must provide written informed consent prior to the conduct of any trial-related procedures.
2. Male or female, 18-65 years of age, inclusive.
3. Diagnosis of moderate or severe opioid use disorder as described (DSM-V).
4. Voluntarily seeking treatment for opioid use disorder.
5. Have not received medication-assisted treatment for opioid use disorder within 60 days prior to randomization.
6. Considered by the Investigator to be a good candidate for BPN treatment, based on medical and psychosocial history.
7. Male or Female subjects of childbearing potential must be willing to use a reliable method of contraception during the entire trial (Screening visit to Follow-up visit)

Exclusion Criteria:

1. Current diagnosis of Acquired Immune Deficiency Syndrome (AIDS).
2. Current diagnosis of chronic pain requiring opioids for treatment.
3. Current DSM-V diagnosis of moderate to severe substance use disorder on any other psychoactive substances other than opioids, caffeine or nicotine (e.g., alcohol, cocaine, sedatives).
4. Pregnant or lactating or planning to become pregnant during the trial.
5. Hypersensitivity or allergy to BPN or other opioids, naloxone or other opioid antagonists, or excipients of CAM2038 or SL BPN.
6. Requires current use of agents that are strong inhibitors or inducers of cytochrome P450 3A4 (CYP3A4) such as some azole antifungals (e.g., ketoconazole), macrolide antibiotics (e.g., clarithromycin), or protease inhibitors (e.g., ritonavir, indinavir, and saquinavir).
7. Subjects with active signs or symptoms of hepatitis and requiring treatment. Subjects with no acute signs of inflammation, and no clinical necessity for therapy will be allowed, at the discretion of the Investigator.
8. Recent history of or current evidence of suicidal ideation or active suicidal behavior as based on the Columbia Suicide Severity Rating Scale (C-SSRS) ("Yes" responses to questions 4 or 5).
9. Any pending legal action that could prohibit participation or compliance in the trial.
10. Exposure to any investigational drug within the 4 weeks prior to Screening.
11. Participants with a history of risk factors of Torsades de Pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome) or an electrocardiogram (ECG) demonstrating a Fridericia's corrected QT interval (QTcF) >450 msec in males and QTcF >470 in females at screening.
12. Aspartate aminotransferase (AST) levels >3 X the upper limit of normal, alanine aminotransferase (ALT) levels >3 X the upper limit of normal, total bilirubin >1.5 X the upper limit of normal, or creatinine >1.5 X upper limit of normal on the Screening laboratory assessments, or other clinically significant laboratory abnormalities, which in the opinion of the Investigator may prevent the subject from safely participating in trial.
13. Significant symptoms, medical conditions, or other circumstances which, in the opinion of the Investigator, would preclude compliance with the protocol, adequate cooperation in the trial or obtaining informed consent, or may prevent the subject from safely participating in trial (including, but not limited to, the risks described as precautions, warnings, and contraindications in the current version of the Investigator's Brochure for CAM2038).
14. Is an employee of the Investigator or the trial site, with direct involvement in the proposed trial or other trials under the direction of the Investigator or trial site, or is a family member of an employee or of the Investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 428 (Actual)
Dates: Start 2015-12; Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Braeburn Pharmaceuticals, Study Chair — Braeburn Pharmaceuticals
Locations (36):
- United States (36):
  - Parkway Medical Center, Birmingham, Alabama
  - Haleyville Clinical Research LLC, Haleyville, Alabama
  - Boyett Health Services Inc, Hamilton, Alabama
  - Synergy East, Lemon Grove, California
  - North County Clinical Research, Oceanside, California
  - Asclepes Research, Panorama City, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Care Practice, San Francisco, California
  - Synergist Research, West Hollywood, California
  - Dr Vijapura and Associates, Jacksonville, Florida
  - Innovative Clinical Research Inc, Lauderhill, Florida
  - TRY Research, Maitland, Florida
  - Tellus Clinical Research, Inc., Miami, Florida
  - Scientific Clinical Research, Inc., North Miami, Florida
  - Professional Research Network of Kansas, LLC, Wichita, Kansas
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Stanley Street Treatment and Resources Inc, Fall River, Massachusetts
  - Novex Clinical Research, New Bedford, Massachusetts
  - Precise Research Centers, Flowood, Mississippi
  - PsychCare Consultants Research, St Louis, Missouri
  - St. Louis Clinical Trials, St Louis, Missouri
  - Wellness and Research Center, Belvidere, New Jersey
  - Comprehensive Clinical Research, Berlin, New Jersey
  - STARS/Columbia University, New York, New York
  - Neuro-Behavioral Clinical Research Center, Canton, Ohio
  - Midwest Clinical Research Center, Dayton, Ohio
  - North Star Medical Research, Middleburg Heights, Ohio
  - Rivus Wellness & Research Institute, Oklahoma City, Oklahoma
  - Frost Medical Group, Conshohocken, Pennsylvania
  - The University of Pennsylvania Health System Treatment Research Center, Philadelphia, Pennsylvania
  - Lincoln Research, Lincoln, Rhode Island
  - Carolina Clinical Trials, Inc, Charleston, South Carolina
  - InSite Clinical Research, Dallas, Texas
  - Aspen Clinical Research, Orem, Utah
  - University of Vermont, Burlington, Vermont
  - Swedish Health Services, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Peterson S, Nunes EV, Lofwall MR, Walsh SL, Tiberg F. Exploring Opioid Use Disorder Outcomes by Quantitative Urinalysis: Post Hoc Analysis of a Phase 3 Randomized Clinical Trial. J Addict Med. 2025 May-Jun 01;19(3):260-267. doi: 10.1097/ADM.0000000000001405. Epub 2024 Dec 4. PMID 39629836
- [Derived] Nunes EV, Comer SD, Lofwall MR, Walsh SL, Peterson S, Tiberg F, Hjelmstrom P, Budilovsky-Kelley NR. Extended-Release Injection vs Sublingual Buprenorphine for Opioid Use Disorder With Fentanyl Use: A Post Hoc Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2024 Jun 3;7(6):e2417377. doi: 10.1001/jamanetworkopen.2024.17377. PMID 38916892
- [Derived] Lofwall MR, Walsh SL, Nunes EV, Bailey GL, Sigmon SC, Kampman KM, Frost M, Tiberg F, Linden M, Sheldon B, Oosman S, Peterson S, Chen M, Kim S. Weekly and Monthly Subcutaneous Buprenorphine Depot Formulations vs Daily Sublingual Buprenorphine With Naloxone for Treatment of Opioid Use Disorder: A Randomized Clinical Trial. JAMA Intern Med. 2018 Jun 1;178(6):764-773. doi: 10.1001/jamainternmed.2018.1052. PMID 29799968

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: SL BPN Tablets + Placebo Subcutaneous (SC) Injections: SL BPN: 2 mg/0.5 mg or 8 mg/2 mg BPN/naloxone tablets administered daily, at doses of 8 mg/2 mg to 32 mg/8 mg per day.
  CAM2038 placebo: 0.16, 0.32, 0.48 and 0.64 mL SC injection administered once weekly or once monthly (matching volumes for CAM2038 q1w and near-matching volumes for CAM2038 q4w).
- Group 2: CAM2038 SC Injections + SL Placebo Tablets: CAM2038 q1w: BPN FluidCrystal® SC injection depot for once weekly administration (50 mg/mL) at doses of 8, 16, 24 and 32 mg (BPN base) (0.16, 0.32, 0.48 or 0.64 mL SC injection).
  CAM2038 q4w: BPN FluidCrystal® SC injection depot for once monthly administration (356 mg/mL) at doses of 64, 96, 128 or 160 mg (BPN base) (0.18, 0.27, 0.36 or 0.45 mL SC injection).
  SL placebo: tablets matching 2 mg/0.5 mg and 8 mg/2 mg SL BPN doses, administered daily
Period: Overall Study
Arm/Group | Group 1: SL BPN Tablets + Placebo Subcutaneous (SC) Injections | Group 2: CAM2038 SC Injections + SL Placebo Tablets
Started | 215 | 213
Completed | 126 | 121
Not Completed | 89 | 92

BASELINE CHARACTERISTICS:
Population: Includes all subjects who were randomized and receiving at least one dose of study drug.
Groups:
- Group 1: SL BP/NX Tablets + Placebo SC Injections: SL BPN/NX: 2 mg/0.5 mg or 8 mg/2 mg BPN/naloxone tablets administered daily, at doses of 8 mg/2 mg to 32 mg/8 mg per day.
  CAM2038 placebo: 0.16, 0.32, 0.48 and 0.64 mL SC injection administered once weekly or once monthly (matching volumes for CAM2038 q1w and near-matching volumes for CAM2038 q4w).
- Total: Total of all reporting groups
Arm/Group | Group 1: SL BP/NX Tablets + Placebo SC Injections | Group 2: CAM2038 SC Injections + SL Placebo Tablets | Total
Number analyzed (Participants) | 215 | 213 | 428
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.0 (10.89) | 38.7 (11.17) | 38.4 (11.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 92 | 165
  Male | 142 | 121 | 263
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 48 | 47 | 95
  White | 164 | 159 | 323
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Hispanic or Latino | 24 | 25 | 49
  Race/Ethnicity: Not Hispanic or Latino | 191 | 188 | 379
BMI [Mean (Standard Deviation); unit: kg/m^2] | 26.2 (5.55) | 25.6 (5.03) | 25.9 (5.30)

OUTCOME MEASURES:

1. Primary Outcome: Response Rate, Denoted by Response Rate (Weeks 1-24).
Description: Response Rate, denoted by response rate (Weeks 1-24). A responder is defined as a subject with at least 33% of urine toxicology results collected during the Phase 1 (4 out of 12 urine samples) and 67% of urine toxicology results collected during Phase 2 (4 out of 6 urine samples) being negative for illicit opioids and self - reported illicit opioid use.
Time Frame: 24 weeks
Population: Includes all subjects who were randomized and receiving at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: SL BP/NX Tablets + Placebo SC Injections | Group 2: CAM2038 SC Injections + SL Placebo Tablets
Number analyzed (Participants) | 215 | 213
Participants
  Responder | 31 | 37
  Non-Responder | 184 | 176
Statistical Analysis 1: Comparison: Group 1: SL BP/NX Tablets + Placebo SC Injections vs Group 2: CAM2038 SC Injections + SL Placebo Tablets; Test type: Non-Inferiority — The p-value was based on the chi square test for non-inferiority with the margin of 10% point; p < 0.001, Chi-squared

2. Secondary Outcome: Cumulative Distribution Function (CDF) of Percentage of Urine Samples Negative for Illicit Opioids
Description: Cumulative distribution function (CDF) of percentage of urine samples negative for illicit opioids comparing CAM2038 to SL BPN/NX as (supported by self-reported opioid use results)
Time Frame: 24 weeks
Population: Includes all subjects who were randomized and receiving at least one dose of study drug.
Measure: Median (Full Range); unit: percentage of negative urine samples
Groups:
- SL BPN Tablets + Placebo Subcutaneous (SC) Injections: SL BPN: 2 mg/0.5 mg or 8 mg/2 mg BPN/naloxone tablets administered daily, at doses of 8 mg/2 mg to 32 mg/8 mg per day.
  CAM2038 placebo: 0.16, 0.32, 0.48 and 0.64 mL SC injection administered once weekly or once monthly (matching volumes for CAM2038 q1w and near-matching volumes for CAM2038 q4w).
Arm/Group | SL BPN Tablets + Placebo Subcutaneous (SC) Injections | Group 2: CAM2038 SC Injections + SL Placebo Tablets
Number analyzed (Participants) | 215 | 213
percentage of negative urine samples
  With Subjects' Self Reported Opioid Use | 0.0 [0.0 to 100.0] | 26.7 [0.0 to 100.0]
  Without Subjects' Self reported Opioid Use | 6.7 [0.0 to 100.0] | 26.7 [0.0 to 100.0]
Statistical Analysis 1: Comparison: SL BPN Tablets + Placebo Subcutaneous (SC) Injections vs Group 2: CAM2038 SC Injections + SL Placebo Tablets; including subject self-reported opioid use; Test type: Superiority; p = 0.004, Wilcoxon Rank-Sum
Statistical Analysis 2: Comparison: SL BPN Tablets + Placebo Subcutaneous (SC) Injections vs Group 2: CAM2038 SC Injections + SL Placebo Tablets; not including self-reported opioid use; Test type: Superiority; p = 0.008, Wilcoxon Rank-Sum

3. Secondary Outcome: Number of Subjects With Sustained Abstinence of Opioid Use
Description: Number of Subjects with Sustained Abstinence of Opioid Use taking SL BPN/NX and CAM2038
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Group 1: SL BPN/NX Tabs+ Placebo Subcutaneous (SC) Injections: SL BPN: 2 mg/0.5 mg or 8 mg/2 mg BPN/naloxone tablets administered daily, at doses of 8 mg/2 mg to 32 mg/8 mg per day.
  CAM2038 placebo: 0.16, 0.32, 0.48 and 0.64 mL SC injection administered once weekly or once monthly (matching volumes for CAM2038 q1w and near-matching volumes for CAM2038 q4w).
Arm/Group | Group 1: SL BPN/NX Tabs+ Placebo Subcutaneous (SC) Injections | Group 2: CAM2038 SC Injections + SL Placebo Tablets
Number analyzed (Participants) | 215 | 213
Participants
  Subjects with sustained abstinence of opioids | 30 | 39
  Subjects without sustained abstinence of opioids | 185 | 174

4. Secondary Outcome: Number of Subjects Remaining in the Study (Retention Rate)
Description: Number of Subjects Remaining in the Study (Retention Rate) on SL BPN/NX and CAM2038
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Group 1: SL BPN/NX Tablets + Placebo SC Injections: SL BPN/NX: 2 mg/0.5 mg or 8 mg/2 mg BPN/naloxone tablets administered daily, at doses of 8 mg/2 mg to 32 mg/8 mg per day.
  CAM2038 placebo: 0.16, 0.32, 0.48 and 0.64 mL SC injection administered once weekly or once monthly (matching volumes for CAM2038 q1w and near-matching volumes for CAM2038 q4w).
Arm/Group | Group 1: SL BPN/NX Tablets + Placebo SC Injections | Group 2: CAM2038 SC Injections + SL Placebo Tablets
Number analyzed (Participants) | 215 | 213
Participants
  Retained | 126 | 121
  Not Retained | 89 | 92
Statistical Analysis 1: Comparison: Group 1: SL BPN/NX Tablets + Placebo SC Injections vs Group 2: CAM2038 SC Injections + SL Placebo Tablets; Test type: Non-Inferiority or Equivalence — The p-value was based on the chi square test for non-inferiority with the margin of 15%; p = 0.006, Chi-squared

ADVERSE EVENTS:
Time Frame: 31 weeks
Groups:
- Group 1: SL BPN/NX Tablets + Placebo SC Injections: SL BPN: 2 mg/0.5 mg or 8 mg/2 mg BPN/naloxone tablets administered daily, at doses of 8 mg/2 mg to 32 mg/8 mg per day.
  CAM2038 placebo: 0.16, 0.32, 0.48 and 0.64 mL SC injection administered once weekly or once monthly (matching volumes for CAM2038 q1w and near-matching volumes for CAM2038 q4w).
Arm/Group | Group 1: SL BPN/NX Tablets + Placebo SC Injections | Group 2: CAM2038 SC Injections + SL Placebo Tablets
All-Cause Mortality (participants affected / at risk) | 0/215 | 1/213
Serious Adverse Events (participants affected / at risk) | 16/215 | 5/213
Other Adverse Events (participants affected / at risk) | 119/215 | 128/213
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: SL BPN/NX Tablets + Placebo SC Injections (N=215) | Group 2: CAM2038 SC Injections + SL Placebo Tablets (N=213)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Acute Hepatitis C (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Localized infection (Infections and infestations) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0)
Accidental Overdose (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Intentional Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bipolar disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Substance-induce mood disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal Ideation (Psychiatric disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Non-cardiac Chest Pain (General disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Chronic Obstructive Pulmonary Disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemophilia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: SL BPN/NX Tablets + Placebo SC Injections (N=215) | Group 2: CAM2038 SC Injections + SL Placebo Tablets (N=213)
Injection site pain (General disorders) | 17 (17) | 19 (19)
Injection site pruritus (General disorders) | 13 (13) | 13 (13)
Injection site erythema (General disorders) | 12 (12) | 12 (12)
Injection site reaction (General disorders) | 7 (7) | 8 (8)
Injection site swelling (General disorders) | 6 (6) | 9 (9)
Injection site induration (General disorders) | 6 (6) | 4 (4)
Injection site inflammation (General disorders) | 8 (8) | 2 (2)
Urinary tract infection (Infections and infestations) | 10 (10) | 11 (11)
Upper respiratory tract infection (Infections and infestations) | 9 (9) | 9 (9)
Cellulitis (Infections and infestations) | 7 (7) | 1 (1)
Constipation (Gastrointestinal disorders) | 16 (16) | 16 (16)
Nausea (Gastrointestinal disorders) | 17 (17) | 15 (15)
Vomiting (Gastrointestinal disorders) | 8 (8) | 9 (9)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 6 (6)
Toothache (Gastrointestinal disorders) | 8 (8) | 3 (3)
Headache (Nervous system disorders) | 17 (17) | 16 (16)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 7 (7)
Back Pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 3 (3)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0)
Insomnia (Psychiatric disorders) | 6 (6) | 12 (12)
Anxiety (Psychiatric disorders) | 7 (7) | 6 (6)
Tachycardia (Cardiac disorders) | 5 (5) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2016-11-04): https://cdn.clinicaltrials.gov/large-docs/84/NCT02651584/SAP_000.pdf
  • Study Protocol (2016-11-03): https://cdn.clinicaltrials.gov/large-docs/84/NCT02651584/Prot_001.pdf